CLINICAL TRIAL: NCT04322890
Title: Treatment Strategies and Survival Outcome for Non-small Cell Lung Cancer With Oncogenic Mutation.
Acronym: PIKACHU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200311
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation; ALK Gene Mutation; ROS1 Gene Mutation; MET Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Erlotinib Hydrochloride; Gefitinib; aflutinib; alectinib; lorlatinib; brigatinib; Crizotinib; entrectinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Drug Therapy; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A: EGFR mutation (Experimental): Lung Cancer with EGFR mutation including EGFR exon19del, exon 21L858R, etc.
  Interventions: Drug: Osimertinib
- Cohort B: ALK fusion (Experimental): Lung Cancer with ALK fusion.
  Interventions: Drug: Alectinib 150 MG
- Cohort C: ROS1 fusion (Experimental): Lung Cancer with ROS1 fusion.
  Interventions: Drug: Crizotinib 250 MG
- Cohort D: MET alterations (Experimental): Lung Cancer with MET alteration including amplification, exon 14 skipping and met fusion etc.
  Interventions: Drug: Savolitinib, Crizotinib.
- Cohort E: RET fusion (Experimental): Lung Cancer with RET fusion.
  Interventions: Drug: Chemotherapy
- Cohort F: KRAS mutation (Experimental): Lung Cancer with KRAS mutation.
  Interventions: Drug: Chemotherapy
- Cohort G: uncommon mutation (Experimental): Cohort G mainly includes all identified lung cancer mutations except EGFR mut, ALK fusion, ROS1 fusion, MET alterations, KRAS mut and RET fusion. These include: BRAF V600E and non-V600E, NRG fusion, NTRK fusion, ERBB2 amp and mut，NRAS mut, MAP2K1 mut，RIT1 mut, RAF1 mut, FGFR fusion, ARAF mut, HRAS mut etc.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Osimertinib — Osimertinib 80mg, po, qd;
  Other Names: Erlotinib, Gefitinib, Furmonertinib, Almonertinib etc.
  Arms: Cohort A: EGFR mutation
Drug: Alectinib 150 MG — Alectinib 600mg, po, qd; Lorlatinib, 100mg, po, qd;
  Other Names: Lorlatinib, Alectinib, Brigatinib, Ceritinib etc.
  Arms: Cohort B: ALK fusion
Drug: Crizotinib 250 MG — Crizotinib 250 MG po bid.
  Other Names: Entrectinib
  Arms: Cohort C: ROS1 fusion
Drug: Savolitinib, Crizotinib. — Savolitinib, 300mg po qd.
  Other Names: Crizotinib
  Arms: Cohort D: MET alterations
Drug: Chemotherapy — 500mg, ivgtt, every 21day.
  Other Names: Pemetrexed, Cisplatin; Pralsetinib etc.
  Arms: Cohort E: RET fusion; Cohort F: KRAS mutation; Cohort G: uncommon mutation

SUMMARY:
The purpose of this study is to assess the Treatment Strategies and Survival Outcome for Non-small Cell Lung Cancer With Oncogenic Mutation.

DETAILED DESCRIPTION:
The purpose of this study is to assess the Treatment Strategies and Survival Outcome for Non-small Cell Lung Cancer With Oncogenic Mutation.

Our study was set up with several group with EGFR mutant, ALK fusion, ROS1 fusion, RET fusion, BRAF mutation, NRG1 fusion, MET alteration, KRAS mutation, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed, Stage IV NSCLC.
4. Oncogenic mutations confirmed by an accredited local laboratory, including EGFR, ALK, ROS1 etc.
5. ECOG 0-1.
6. Predicted survival ≥ 12 weeks.
7. Adequate bone marrow hematopoiesis and organ function
8. Presence of measurable lesions according to RECIST 1.1.

Exclusion Criteria:

The patient did not match from the Inclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated with target treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | To assess overall survival, define as first dose to the death of the subject due to any cause up to 5 years
  To assess overall survival, define as first dose to the death of the subject due to any cause
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated with target treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause.
Adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0
Patient reported outcome (PRO) | To assess overall survival, define as first dose to the death of the subject due to any cause up to 5 years
  Patient reported outcome defined as the quality of life during the whole process treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China